CLINICAL TRIAL: NCT07154901
Title: A Single-Dose, Non-Randomised, Open-Label, Parallel-Group Study to Investigate the Effects of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of Opemalirsen (AZD2373)
Brief Title: Investigation of the Effects of Renal Impairment on the Pharmacokinetics, Safety, and Tolerability of Opemalirsen (AZD2373)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D6800C00006
Record Dates: First submitted 2025-07-28; First posted 2025-09-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Renal Impairment
Keywords: Renal impairment; AZD2373; Pharmacokinetics; Severe; Mild; Moderate; Matched Healthy Controls; opemalirsen
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to the following groups based on BSA-adjusted eGFR at screening using the creatinine-based CKD-EPI (2021) race-free estimation of eGFR:
  * Part 1:
    * Group 1: Participants with normal renal function (eGFR ≥ 90 mL/min; n = 8 to 20 participants)
    * Group 2: Participants with severe renal impairment not on dialysis (eGFR < 30 mL/min; n = 8 to 10 participants)
  * Part 2 (Optional):
    * Group 3: Participants with moderate renal impairment (eGFR ≥ 30 mL/min to < 60 mL/min; n = 8 to 10 participants)
    * Group 4: Participants with mild renal impairment (eGFR ≥ 60 mL/min to < 90 mL/min; n = 8 to 10 participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Healthy participants will receive a single subcutaneous injection of AZD2373.
  Interventions: Drug: Opemalirsen (AZD2373)
- Group 2 (Experimental): Severe renal impairment participants will receive a single subcutaneous injection of AZD2373.
  Interventions: Drug: Opemalirsen (AZD2373)
- Group 3 (Experimental): Moderate renal impairment participants will receive a single subcutaneous injection of AZD2373
  Interventions: Drug: Opemalirsen (AZD2373)
- Group 4 (Experimental): Mild renal impairment participants will receive a single subcutaneous injection of AZD2373
  Interventions: Drug: Opemalirsen (AZD2373)

INTERVENTIONS:
Drug: Opemalirsen (AZD2373) — Single, subcutaneous injection of AZD2373

SUMMARY:
This study is being conducted to investigate the PK, safety, and tolerability of opemalirsen in participants with renal impairment, compared to participants with normal renal function.

DETAILED DESCRIPTION:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study, that will be conducted in 2 parts, to examine the PK, safety, and tolerability of opemalirsen in male and female participants with severe renal impairment to matched participants with normal renal function; and, if necessary, participants with mild and moderate renal impairment to matched participants with normal renal function.

Potential participants will be screened to assess their eligibility to enter the study within 28 days prior to first dose administration. Participants will be assigned to the following groups based on BSA-adjusted eGFR at screening using the creatinine-based CKD-EPI (2021) race-free estimation of eGFR:

* Part 1:

  * Group 1: Participants with normal renal function (eGFR ≥ 90 mL/min; n = 8 to 20 participants)
  * Group 2: Participants with severe renal impairment not on dialysis (eGFR < 30 mL/min; n = 8 to 10 participants)
* Part 2 (Optional):

  * Group 3: Participants with moderate renal impairment (eGFR ≥ 30 mL/min to < 60 mL/min; n = 8 to 10 participants)
  * Group 4: Participants with mild renal impairment (eGFR ≥ 60 mL/min to < 90 mL/min; n = 8 to 10 participants)

If the data from Part 1 demonstrate that severe renal impairment does not alter PK of opemalirsen to an extent which would warrant dose adjustment, then Part 2 will not be pursued. If the PK data of the study support a dosage adjustment in patients with severe renal impairment, then participants will be enrolled Group 3 and/or Group 4 in Part 2. Additional participants may be enrolled in Group 1 (not exceeding n = 20) and dosed in parallel with Part 2, if required, to match participants in Groups 3 and/or 4.

Each matched participant with normal renal function (Group 1) enrolled in the study will be demographically matched by sex, age (± 10 years), and BMI (± 20%), data obtained at screening, to an enrolled participant with renal impairment. Participants with normal renal function cannot be matched to more than one participant with renal impairment within an impairment group; however, participants with normal renal function may be matched to

1 participant from more than 1 renal impairment group.

Eligible participants will be admitted to the study site on Day -1. On Day 1, participants will receive a single SC injection of opemalirsen. Participants will be confined to the study site until Day 3 and will return for follow-up visits 1, 2, 3, and 8 weeks post-dose.

Serial PK (venous) blood samples and urine samples will be collected up to 48 hours post-dose (Day 3) for the measurement of opemalirsen in plasma and urine. Additional blood samples will be collected the follow-up visits 1, 2, and 3 weeks post-dose for the measurement of opemalirsen in plasma. Adverse events and serious adverse events will be recorded and physical examinations, 12-lead electrocardiograms, vital sign measurements, and clinical laboratory tests will be performed to assess safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. Participant must be 18 to 80 years of age, inclusive, at the time of signing the informed consent. Type of Participant and Disease Characteristics For all participants, BSA-adjusted eGFR will be determined by the local laboratory, calculated based on serum creatinine using the CKD-EPI equation (see Section 4.1).

   Healthy matched control participants only (Group 1):
2. Participant must be medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, or 12-lead ECGs, as deemed by the investigator at screening and Day -1.
3. Have an eGFR of ≥ 90 mL/min determined at screening.

Participants with renal impairment only (Group 2 and optional Groups 3 and 4):

4 Diagnosis of chronic kidney disease with stable renal function in the 3 months prior to dosing, as determined by the investigator, based on medical history or eGFR, and not requiring dialysis. 5 Participants with renal impairment, as follows, based on CKD-EPI equation (BSA-adjusted eGFR) at screening:

1. Group 2: have severe renal impairment (eGFR < 30 mL/min), not requiring dialysis.
2. Group 3 (optional): have moderate renal impairment (eGFR ≥ 30 to < 60 mL/min)
3. Group 4 (optional): have mild renal impairment (eGFR ≥ 60 to < 90 mL/min) 6 Participants on angiotensin-converting enzyme inhibitors/angiotensin II receptor blockers, beta-blocker, diuretics, or on any other cardiorenal relevant treatment should be on a stable dose for at least 2 weeks prior to screening. Weight 7 Body weight of at least 50 kg and body mass index (BMI) within the range 18 to 40 kg/m2 (inclusive). Sex and Contraceptive/Barrier Requirements 8 Male and/or female, assigned at birth, inclusive of all gender identities. 9 Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

(a) Male participants must agree to the following contraception guidance for the duration of the study (from the time of study intervention administration) until 3 months after discharge: (i) Non-sterilised male participants should avoid fathering a child by either true abstinence or by using (together with their female partner/spouse) a highly effective contraception form of birth control in combination with a barrier method, starting from the time of study intervention administration until 3 months after discharge. Acceptable methods of preventing pregnancy include birth control pills, injections, implants, or patches, IUDs, tubal ligation/occlusion, and vasectomy. (ii) Male participants who have been sterilised are required to use one barrier method of contraception (condom) from the time of study intervention administration until after discharge. A barrier method is not necessary if the female partner is sterilised. (iii) Male participants should not donate sperm from the time of study intervention administration until 3 months after discharge. (b) Female participants: must not be pregnant and must have a negative pregnancy test at screening (all female participants) and check-in (WOCBP) and must not be lactating.

Women of Childbearing Potential (WOCBP): A woman is considered of childbearing potential if she is capable of conceiving. While this is typically the case following menarche and up until she becomes post-menopausal, adolescents can ovulate prior to first menarche, and women with irregular menses may also be fertile. Women Not of Childbearing Potential (WNOCBP): Females not of childbearing potential are defined as females who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are post-menopausal. Females will be considered post-menopausal if they have been amenorrhoeic for 12 months prior to the planned date of dose administration without an alternative medical cause. The following age-specific requirements apply:

* Females < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
* Females ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment. (i) Female participants should be stable on the chosen method of contraception for a minimum of 3 months before entering the study. (ii) Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Females of childbearing potential who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control, as defined below, throughout the study and until at least 3 months after discharge. Cessation of contraception after this point should be discussed with a responsible physician. Note: contraception is not required for female participants of non-childbearing potential.

  * Highly effective birth control methods include:

    * Non-hormonal • Total sexual abstinence provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments) • a vasectomised partner (confirmed absence of sperm in semen) • bilateral tubal occlusion

      • intrauterine device (copper)
    * Hormonal contraceptives associated with inhibition of ovulation levonorgestrel intrauterine system • medroxyprogesterone injections • combined Oral or transdermal contraceptives (ethinyl estradiol plus progestin) • intravaginal device (eg, EE and etonogestrel) The following are not acceptable methods of contraception: female condom, periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea.

Exclusion Criteria:

* Medical Conditions

All participants:

1. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the investigator, at screening or Day -1, or history of hypersensitivity to drugs with a similar chemical structure or class to opemalirsen.
2. History of any major surgical procedure within 30 days prior to study intervention.
3. Judgement by the investigator that the participant should not participate in the study if they have any ongoing or recent (ie, during the screening period) minor medical complaints that may interfere with the interpretation of study data or if they are considered unlikely to comply with study procedures, restrictions, and requirements.
4. Liver disease (non-alcoholic and alcoholic steatohepatitis; drug-induced, viral, or autoimmune hepatitis; primary biliary cirrhosis; primary sclerosing cholangitis; hemochromatosis; alpha-1 antitrypsin deficiency; Wilson's disease) including positive results for hepatitis B surface antigen, hepatitis B core antibody or hepatitis C virus antibody.
5. History of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy, or variceal bleeding.
6. QTcF > 470 ms in participants without bundle branch block and > 480 ms in participants with bundle branch block.
7. Any of the following out of range laboratory values:

   1. ALT or AST > 1.5 × ULN
   2. TBL > ULN (an isolated increase in TBL in participants with Gilbert syndrome is not a reason for exclusion)
   3. INR > 1.2, unless related to therapeutic anticoagulation
   4. APTT ≥ 1.3 × normal, unless related to therapeutic anticoagulation
   5. HbA1c ≥ 10%
8. Positive test for human immunodeficiency virus at screening.
9. Known history of drug or alcohol abuse within 1 year of screening.

   Healthy matched control participants only (Group 1):
10. Any clinically significant disease or disorder (eg, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal including bone fractures, endocrine including adrenal insufficiency, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the investigator, may put the participant at risk because of participation in the study, influence the results of the study, or affect the participant's ability to participate in the study.
11. Abnormal resting vital signs (after resting for 10 minutes) of supine BP > 150 mmHg or < 90 mmHg systolic or > 95 mmHg or < 50 mmHg diastolic or supine pulse rate ≥ 100 bpm or ≤ 45 bpm. Note: the blood pressure values will be based on the average of the 3 measurements.

    Participants with renal impairment only (Group 2 and optional Groups 3 and 4):
12. Evidence of rapidly deteriorating renal function.
13. Presence of unstable medical (eg, diabetes) or psychological conditions which, in the opinion of the investigator, would compromise the participant's safety or successful participation in this study.
14. Renal transplant patients, that is, participants that have received a kidney transplant or participants waiting for organ transplant scheduled to occur during the study, and those with a history of acute kidney injury occurring within 3 months prior to screening.
15. Abnormal resting vital signs (after resting for 10 minutes) of supine BP > 180 mmHg or < 110 mmHg systolic or > 110 mmHg or < 60 mmHg diastolic or supine pulse rate ≥ 100 bpm or ≤ 40 bpm. Note: the blood pressure values will be based on the average of the 3 measurements.

    Prior/Concomitant Therapy

    Healthy matched control participants only (Group 1):
16. Use of any prescription or non-prescription drugs (including vitamins, recreational drugs, and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before study intervention, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study.

    Participants with renal impairment only (Group 2 and optional Groups 3 and 4):
17. Use of concurrent medication, which affect creatinine clearance such as cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine, quinine within 7 days prior to Day -1.

    Prior/Concurrent Clinical Study Experience

    All participants:
18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days of study intervention in this study or, if known, 5 half-lives from last dose in the previous study to study intervention in this study, whichever is longest.
19. Previous enrolment in the present study. Note: participants consented and screened, but not receiving study intervention in this study or a previous Phase I study, are not excluded. Other Exclusions

    All participants:
20. Positive screen for drugs of abuse (unless participant has renal impairment and positive screen is due to medication[s] prescribed by physician) and/or alcohol test at screening or Day -1; a positive result for tetrahydrocannabinol and/or cannabinoids is not considered exclusionary.
21. Receipt of blood products within 2 months prior to Day -1, plasma or platelets donation within 1 month prior to Day -1, or any blood donation/blood loss > 500 mL within

3 months prior to Day -1. 22 Involvement of any AstraZeneca or clinical unit employee or their close relatives.

23 Vulnerable participants, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order. 24 Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
AUCinf | Pre-dose to 3 weeks post dose
  Area under the concentration-time curve from zero to infinity
AUClast | Pre-dose to 3 weeks post-dose
  Area under the concentration-time curve from zero to the last measurable concentration
Cmax | Pre-dose to 3 weeks post-dose
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Tmax | Pre-dose to 3 weeks post-dose
  Time to reach maximum observed plasma concentration
t1/2λz | Pre-dose to 3 weeks post-dose
  Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve
CL/F | Pre-dose to 3 weeks post-dose
  Apparent total body clearance of drug from plasma after extravascular administration
Vz/F | Pre-dose to 3 weeks post-dose
  Apparent volume of distribution during the terminal phase after extravascular administration
Fu | Pre-dose to 3 weeks post-dose
  Fraction unbound
CLr | Pre-dose to 3 weeks post-dose
  Renal clearance of the drug from plasma
Ae | Pre-dose to 3 weeks post-dose
  Cumulative amount of unchanged drug excreted into the urine
fe | Pre-dose to 3 weeks post-dose
  Fraction of the drug excreted into the urine

OTHER OUTCOMES:
Number of Participants with Abnormal AEs and SAEs | Screening to Day 57
  Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home